CLINICAL TRIAL: NCT04740541
Title: Determination of Threonine Requirement in Adult Males With Crohn's Disease Using the Indicator Amino Acid Oxidation (IAAO) Methodology
Brief Title: Threonine Requirement in Adult Males With Crohn's Disease Using IAAO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: MOUNT SINAI HOSPITAL (Other)
Responsible Party: Principal Investigator, Glenda Courtney-Martin, Project Investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000062867
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Crohn Disease; IBD
Keywords: indicator amino acid oxidation; threonine requirement
MeSH Terms: conditions — Crohn Disease | interventions — Eating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Threonine Requirement in CD Patients (Experimental): Males aged 18 - 49 with stable Crohn's disease will be seen for pre-study They will be studied up to 5 times for different levels of threonine intakes.
  Interventions: Other: Dietary Intakes (Reference protein drinks (Scandishake, Solcarb, Beneprotein) and cookies)

INTERVENTIONS:
Other: Dietary Intakes (Reference protein drinks (Scandishake, Solcarb, Beneprotein) and cookies) — Reference protein drinks (Scandishake, Solcarb, Beneprotein) and cookies to meet nutritional requirements, 5 levels of threonine intakes

SUMMARY:
The goal of the current study is to measure the requirement for threonine in patients with CD using the IAAO method and compare the requirement to previously determined threonine requirement estimated in young adults using the IAAO technique. It is hypothesize that the requirement for threonine in patients with CD will be higher than the threonine requirement previously determined in young adults using the IAAO method. Up to 10 clinically stable patients with CD will be recruited from the IBD Clinic at Mt. Sinai Hospital, Toronto, and subsequently followed up at the Clinical Research Center (CRC), The Hospital for Sick Children (SickKids), Toronto, Canada. Before the study begins, the participants will be required to visit the CRC (Room 5500 Hill Wing, The Hospital for Sick Children) for a pre-study assessment of their height, weight, fat mass, fat free mass, resting metabolic rate and medical history. These assessments will take about 3 hours to complete. They will need to have been fasted for 10 hours prior to the pre-study assessment. The pre-study assessment is needed to calculate their dietary requirements for the study, and to assess health status. After signing the consent form, the subjects will complete the screening procedures (height, weight, fasting blood sample and medical history questionnaire, BIA, Skinfold and calorimetry).

Each study will consist of a 2-day adaptation period to a prescribed diet in accordance with the energy requirement of the subject and 1-study day. The diet will provide an adequate amount of protein, of 1 g protein/kg/d. The 2-day adaptation period is to allow the body to adapt to an adequate amount of protein as it has been shown that protein kinetics is altered without it.

Dietary intakes during this time will be provided in the form of lactose-free milk shakes (Scandishake) with added carbohydrate (SolCarb) and protein (beneprotein) to meet the subjects' requirement.

Following the 2 days of adaptation is the study day where threonine intake will be randomly assigned and phenylalanine (Phe) kinetics will be measured with the use of isotopically labelled Phe. On this day, VCO2 will be measured by calorimetry immediately after the 5th meal for a period of 20 minutes.

On the study day (3rd day of each 3-day period), the diet will be provided as 8 hourly isocaloric, isonitrogenous meals made up of a flavored liquid formula and protein free cookies developed for use in amino acid kinetic studies. Each meal will represent 1/12th of the subject's total daily requirements. The nitrogen (protein) content of the diet will be provided in the form of a crystalline amino acid mixture based on the amino acid composition of egg protein.

* A daily multivitamin supplement will be provided during the study period.
* No other food or beverages will be consumed on the adaptation days except water, 1 cup clear tea, or 1 cup clear coffee.
* During the 8-hr study day, no other food or drink will be consumed except water.
* Urine and breath samples will be collected at baseline and at isotopic steady state.
* Breath samples will be collected simultaneously with urine samples.
* Five baseline breath samples will be collected 60, 45, 30, 15 min, and just before the tracer protocol begins.
* Three baseline urine samples will be collected 60, 30 min, and just before the tracer protocol begins.
* Four plateau breath samples will be collected every 15 minutes 2.5 h after the tracer protocol begins.
* Three plateau breath samples will be collected every 30 minutes 2.5 h after the tracer protocol begin
* Breath samples will be collected with subjects breathing into an Exetainers plastic tube and samples will be stored in pre-evacuated glass tubes at room temperature until analysis.
* Urine samples will be collected in Eppendorf tubes and stored at - 20 º C until analyzed for 1-13C phenylalanine enrichment.
* The rate of CO2 production (VCO2) will be measured on each testing day using a ventilated hood indirect calorimeter at meal 5 to quantify 13CO2 excretion in breath.

Subjects can choose to withdraw from the study at any time and for any reason, based on his/her individual judgment. In particular, if a subject is unable to tolerate the diet, whether it is regards to taste, loose stools or constipated stools, he/she has the right to withdraw at any time during the study.

DETAILED DESCRIPTION:
BACKGROUND The current Dietary Reference Intake (DRI) recommendations for essential amino acid requirements are based on recommendations for young healthy adults and have not been directly determined in patients with Crohn's disease. Protein and amino acids are key components of our diet. Having defined the requirement of the essential amino acid, Threonine in healthy adults using the IAAO, the investigators are now in an ideal position to define the needs in vulnerable populations, such as patients with chronic inflammatory conditions, such as Crohn's disease (CD).

Studies in animals suggest an increase in the threonine requirement in Crohn's and colitis models. If this is also true in humans, knowledge of the threonine requirement in patients with IBD could provide valuable information for improvement in medical nutritional management of this patient population. Improved medical nutrition therapy could likely shorten recovery time and/or increase the period of remission in patients with IBD.

Method:

Indicator Amino Acid Oxidation

Hypothesis:

It is hypothesized that the requirement for threonine in patients with CD will be higher than the threonine requirement previously determined in young adults using the IAAO method (19 mg/kg/d).

Objectives:

1. To determine the requirement for threonine in patients with CD using the IAAO technique; by measuring the oxidation of L-[1-13 C] phenylalanine to 13 CO 2 [F 13 CO 2] in response to graded intakes of leucine.
2. To compare, on the basis of body weight and fat-free mass, the requirement derived from this study to the requirement of threonine determined previously in young adults by the IAAO method.

Subjects:

Up to 10 clinically stable patients with CD will be recruited from the IBD Clinic at Mt. Sinai Hospital, Toronto, who will be identified by Dr. Mark Silverberg for this study and subsequently followed up at the Clinical Research Center (CRC), The Hospital for Sick Children (SickKids), Toronto, Canada. Before the study begins, the participants will be required to visit the CRC (Room 5500 Hill Wing, The Hospital for Sick Children) for a pre-study assessment of their height, weight, fat mass, fat free mass, resting metabolic rate and medical history. These assessments will take about 3 hours to complete. They will need to have been fasted for 10 hours prior to the pre-study assessment. We need the pre-study assessment to calculate their dietary requirements for the study, and to assess health status.

After signing the consent form, the subjects will complete the screening procedures (height, weight, fasting blood sample and medical history questionnaire, BIA, Skinfold and calorimetry).

* The voluntaries will receive financial compensation for the costs incurred while participating in the study.
* All procedures in the study will be approved by the Research Ethics Board at SickKids.

Experimental Design:

The experimental design will be based on the minimally invasive IAAO model for collecting breath and urine, instead of blood during the study day. A maximum total of 50 IAAO studies will be carried out to determine the requirement for threonine in patients with CD. Up to 10 male patients with CD will be recruited. Each subject will be studied for at least 2 intake levels and up to at a maximum of 5 different intake levels of threonine. Each level of intake will be randomly assigned to subjects.

At the pre-study assessment, the subject's resting energy expenditure (REE) will be measured by continuous, open-circuit indirect calorimetry, and body composition will be measured by skinfold thickness and bioelectrical impedance analysis (BIA). Subjects will also be weighed at the pre-study assessment and at the start of each IAAO study day to ensure accurate prescription of diets and isotopes, and to confirm weight maintenance throughout the study.

Each study will consist of a 2-day adaptation period to a prescribed diet in accordance with the energy requirement of the subject and 1-study day. The diet will provide an adequate amount of protein, of 1 g protein∙kg-1∙d-1. The 2-day adaptation period is to allow the body to adapt to an adequate amount of protein as it has been shown that protein kinetics is altered without it. Following the 2 days of adaptation is the study day where threonine intake will be randomly assigned and phenylalanine (Phe) kinetics will be measured with the use of L-[1-13C]Phe. On this day, VCO2 will be measured by calorimetry immediately after the 5th meal for a period of 20 minutes.

Dietary Intake and Experimental Diet:

3-day protocol

* On days 1 and 2, the subject will consume an adaptation diet and on the 3rd day participate in an 8-hour testing period. Each 3-day protocol will be separated by at least one week (wash-out period).
* Dietary intakes during the 2-day adaptation period before the day 3 IAAO study will be provided in the form of lactose-free milk shakes (Scandishake) with added carbohydrate (SolCarb) and protein (beneprotein) to meet the subjects' requirement. The protein will be provided from the scandishake as milk protein (casein and whey) and providing 1g.kg-1.day-1 protein intake. Total calories will be provided as resting energy expenditure (REE) measure by indirect calorimetry and multiplied by 1.7. On the adaptation days, the diet will be provided as four isonitrogenous, isocaloric meals spread evenly throughout the day.
* On the study day (3rd day of each 3-day period), the diet will be provided as 8 hourly isocaloric, isonitrogenous meals made up of a flavored liquid formula and protein free cookies developed for use in amino acid kinetic studies. Each meal will represent 1/12th of the subject's total daily requirements. The nitrogen (protein) content of the diet will be provided in the form of a crystalline amino acid mixture based on the amino acid composition of egg protein. The energy intake on the study day will be provided as REE x 1.5.
* Tyrosine will be provided in excess at 40 mg/kg/day
* Phenylalanine will be provided at a constant intake of 20mg/kg/d.
* Threonine will be provided at graded intakes ranging from 3-45 mg/kg/d and alanine levels will be adjusted to balance the changing levels of leucine and ensure formulas are isonitrogenous.
* A daily multivitamin supplement will be provided during the study period.
* No other food or beverages will be consumed on the adaptation days except water, 1 cup clear tea, or 1cup clear coffee.
* During the 8-hr study day, no other food or drink will be consumed except water.

Study Day

* The study day diet will be divided into 8 isonitrogenous, isocaloric meals each representing one-twelfth of the total subject´s daily requirements.
* On the morning of each study day, the subject will consume 4 of the hourly meals at home and then visit the research laboratory. The subject will then start to consume the remaining 4 out of the 8 isocaloric meals at hourly intervals.
* Up to 5 dietary threonine intake levels will be tested in random order as mentioned under "experimental design".
* 1-13C phenylalanine will be given as the tracer in the 5th meal and continue to be administered with the remaining meals.

Body-composition measurements

• Body composition will be determined by bioelectrical impedance analysis (BIA and multiple skin fold-thickness measurements at the beginning of study during the pre-study assessment. Four Skinfold thicknesses (triceps, biceps, subscapular, and suprailiac) will be measured to obtain estimates of fat mass. BIA will be performed by using a fixed-frequency analyzer (50 kHz; BIA model 101A: RJL Systems). Equations described previously will be used to calculate FFM.

Isotope Infusion Protocol:

* 1-13C phenylalanine will be used as the isotope. Oral priming dose of 0.66 mg/kg will be administered with the fifth meal, and an hourly oral dose of 1.2 mg/kg/d will begin simultaneously and continue for 3 hrs with meals 6, 7 and 8. A total of 4 isotopic doses are given to ensure background 13CO2 in breath reaches equilibration
* At the same time which the priming dose of L-[13C]phe is administered, an oral priming dose of 0.176 mg/kg of bicarbonate (NaH13CO3) will also be given
* The amount of phenylalanine given as the isotope on the study day will be subtracted from dietary phenylalanine to maintain the total dietary intake at 20 mg Phe /kg/d
* Tyrosine intake will be maintained at 40 mg∙kg-1∙d-1 to ensure an excess of tyrosine
* Breath and urine samples are collected periodically before and after the tracers are consumed

Sample Collection:

* Urine and breath samples will be collected at baseline and at isotopic steady state.
* Breath samples will be collected simultaneously with urine samples.
* Five baseline breath samples will be collected 60, 45, 30, 15 min, and just before the tracer protocol begins.
* Three baseline urine samples will be collected 60, 30 min, and just before the tracer protocol begins.
* Four plateau breath samples will be collected every 15 minutes 2.5 h after the tracer protocol begins.
* Three plateau breath samples will be collected every 30 minutes 2.5 h after the tracer protocol begin
* Breath samples will be collected with subjects breathing into an Exetainers plastic tube and samples will be stored in pre-evacuated glass tubes at room temperature until analysis.
* Urine samples will be collected in Eppendorf tubes and stored at - 20 º C until analyzed for 1-13C phenylalanine enrichment.
* The rate of CO2 production (VCO2) will be measured on each testing day using a ventilated hood indirect calorimeter at meal 5 to quantify 13CO2 excretion in breath.

Sample Analysis.

* Breath: expired 13 CO2 enrichment will be measured by continuous flow isotope ratio mass spectrometer (IRMS).
* Urinary 1-13C phenylalanine enrichment will be analyzed by gas chromatography tandem mass spectrometry (LC-MS-MS).

Estimation of Isotopic Kinetics Whole-body phenylalanine flux will be calculated as previously described according to the stochastic model of Matthews et al. Isotopic steady state in the tracer enrichment at baseline and plateau will be represented as the unchanging values of L-[1-13C]phenylalanine in urine and 13CO2 in breath.

Phenylalanine flux (umol/kg/h) will be calculated from the dilution of orally administered 13C-phenylalanine into the metabolic pool (at steady state) by using enrichment of 13C- phenylalanine in urine. The rate of appearance of 13CO2 in breath (F13CO2 umol/kg/h) after the oxidation of ingested 13C-phenylalanine will be calculated according to the model of Matthews et al., by using a factor of 0.82 to account for carbon dioxide retained in the body's bicarbonate pool. The rate of phenylalanine oxidation (umol/kg/h) will be calculated from F13CO2 and urinary 13C-phenylalanine enrichment.

Statistical Analysis

A paired t test will be used to test for: differences in FFM and percentage of body fat; differences in the two body-composition methods of BIA and skinfold. ANOVA will be used to test for differences among the various estimates of body composition (fat and FFM), and correlation analysis will be performed to test for associations

Threonine intakes will be completely randomized within subjects, with the amount of threonine intake serving as the main treatment effect. The effect of threonine on phenylalanine flux, oxidation, and F13CO2 will be tested by using a mixed linear model with subject as a random variable (PROC MIXED) by using SAS. Differences between individual fluxes will be compared by ANOVA, with post hoc analysis using the Bonferroni multiple-comparisons test.

Threonine requirement will be determined by applying a biphasic linear regression crossover analysis to determine the breakpoint (EAR) and subsequently calculate the 95% CI. The mean threonine requirement will be estimated by applying a nonlinear mixed-effects model (PROC NLMIXED; SAS Institute) to the oxidation and F13CO2 data. Observations within subjects will be regarded as statistically depended.

ELIGIBILITY:
Inclusion Criteria:

* Male 18 - 49 years of age
* Having obtained his (or his legal representative's) written informed consent
* Evidence of ileal and or colon inflammatory involvement and clinically stable disease state and HBI ≤ 8
* Evidence of some active disease based on history of elevated CRP or parameters of active mucosal
* No evidence of intestinal strictures that may affect the subjects' ability to consume a normal diet
* Have maintained a stable weight for at least 3 months and not on enteral feed via tube
* Willingness to participate in the study and completed the screening procedures (height, weight, fasting blood sample and medical history questionnaire) and willingness to consume the diet provided

Exclusion Criteria:

* Uncontrolled inflammation which will likely require surgery or escalation of therapy in the next 4 weeks
* Concomitant treatment: corticosteroid > 20 mg/day
* Subjects without any evidence of inflammatory activity
* On medications known to affect protein and amino acid metabolism (steroids)
* Recent significant weight loss
* Individual on weight reducing diets
* Inability to tolerate the diet
* Subjects who cannot be expected to comply with the study procedures
* Significant coffee consumption of more than 2 cups/day
* Significant alcohol consumption of more than one drink/day

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Requirement of Threonine in Adult Males with Crohn's Disease | 1 - 6 months
  Apply IAAO method to determine the DRI for Threonine in CD patients

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Courtney-Martin, PhD, RD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided